CLINICAL TRIAL: NCT06552910
Title: Diabetic Foot Amputations: A Comprehensive Review of Anesthetic Procedures and Outcomes
Brief Title: Analyzing Anesthetic Techniques in Diabetic Foot Amputation
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, semih başkan, Associate Professor, Ankara City Hospital Bilkent
Other Study IDs: SMH1
Record Dates: First submitted 2024-07-22; First posted 2024-08-14 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Foot; Amputation, Surgical
Keywords: Diabetic Foot; Nerve Block; Diabetes Complications; Amputation, Surgical
MeSH Terms: conditions — Diabetic Foot; Diabetes Complications | interventions — Nerve Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group/Cohort 1: Label: Peripheral Nerve Block Description: Injection of anesthetic near specific nerves to block sensation in a particular area of the body.
  Interventions: Procedure: Nerve Block

INTERVENTIONS:
Procedure: Nerve Block — Since this study was conducted retrospectively, the choice of anesthesia method was made based on our own experience. For every patient undergoing LEA under PNB, a popliteal sciatic nerve block was carried out. A saphenous nerve block was also carried out if the procedure was on a level that was close to the metatarsal bone. In some circumstances (distal surgery, such as the metatarsal bone), a sensory block on the surgical site was tried following the popliteal sciatic nerve block to demonstrate that the saphenous nerve's anatomic abnormalities required an additional saphenous nerve block. The related block was later carried out, if needed. Under ultrasound guidance, every PNB was finished.

SUMMARY:
Diabetic Foot Amputations: A Comprehensive Review of Anesthetic Procedures and Outcomes

Introduction:

Diabetic foot is a severe complication of diabetes, often resulting in ulceration, osteomyelitis, and gangrene. Amputation or surgical debridement is the standard treatment for advanced cases. The study aims to evaluate the outcomes of different anesthetic techniques in diabetic foot amputation, specifically comparing peripheral nerve block (PNB) and general anesthesia.

Objective:

To assess the impact of anesthetic procedures on outcomes in diabetic foot amputation cases using inpatient data. The hypothesis is that PNB will result in fewer postoperative complications than general anesthesia-primary outcome: 30-day mortality; secondary outcomes: composite morbidity and hospital discharge duration.

Materials and Methods:

This retrospective chart review will analyze medical records of patients with diabetic foot at Ankara Bilkent City Hospital from 2021 to 2023. Inclusion criteria: patients who underwent toe, ankle, or foot amputations. Exclusion criteria: patients under 18, amputations for non-diabetic reasons, and insufficient medical data. Data will include patient demographics, preoperative medications, comorbidities, and surgical details. Major complications, secondary outcomes, and mortality will be primary measures.

Statistical Analysis:

Descriptive statistics will summarize patient characteristics. Chi-square and Student t-tests will analyze associations between anesthesia type and postoperative outcomes. Kaplan-Meier survival analysis will compare hospital stay durations. Logistic regression will adjust for confounders and assess the impact of anesthetics on complications. Results will be significant at p < 0.05.

DETAILED DESCRIPTION:
Diabetic Foot Amputations: A Comprehensive Review of Anesthetic Procedures and Outcomes Introduction Diabetic foot is a clinical manifestation of diabetes with a wide range of symptoms, including ulceration, osteomyelitis, osteoarticular destruction, and gangrene, as a consequence of advanced disease. Some cases of diabetic foot present general indications for amputation, including dead limbs, threat to the patient's life, pain, loss of function, or nuisance. Surgical debridement or amputation is the standard treatment for this condition. Multiple debridement operations, however, have been shown in recent research to considerably improve wound healing rates, making them a potential therapeutic alternative. The majority of patients with diabetic foot ulcers are older, have had diabetes for a longer period, have numerous organ problems, and at least one comorbid ailment.

As neuraxial anesthesia, a type of regional anesthetic, does not require positive mechanical breathing and offers superior pain management, less surgical stress response, and enhanced blood flow, it should theoretically result in a better prognosis than general anesthesia. However, due to the increased incidence of macrovascular complications such as peripheral artery occlusive disease, cerebrovascular disease, and coronary heart disease in patients undergoing diabetic foot amputation, prophylactic or therapeutic anticoagulation is necessary. On the other hand, peripheral nerve block (PNB) shares many theoretical advantages of regional anesthesia and can be beneficial in these cases.

The goal of the research is to assess the outcomes of anesthetic procedures carried out in diabetic foot amputation cases using data from an inpatient database. The hypothesis is that peripheral nerve block will be less likely than general anesthesia to cause postoperative complications. The primary outcome is 30-day mortality following lower extremity amputation; secondary outcomes include composite morbidity from potentially fatal sequelae and hospital discharge duration.

Materials and Methods This study will be conducted using a retrospective chart review method. The study will utilize data from the medical records of patients. Medical data from patients with diabetic foot at Ankara Bilkent City Hospital between 2021 and 2023 will be included in the study. These patients will include those who have toe, ankle, or foot amputations. This research will encompass all individuals who had surgery during this time. Patients with diabetic feet who had their feet, ankles, or toes amputated will meet the inclusion criteria. Exclusion criteria will include those under the age of 18, those whose amputations were performed for reasons other than diabetic foot, and those with insufficient medical data.

Since this study will be conducted retrospectively, the choice of anesthesia method was based on clinical experience.

Using the hospital information management system, patients' medical records will be examined retrospectively. Baseline patient demographic data will include age, sex, height, weight, body mass index, nature of the procedure, smoking status, and American Society of Anesthesiologists physical status classification. Preoperative medication records will be gathered, including beta-blockers, calcium channel blockers, insulin, renin-angiotensin system antagonists, anticoagulant or antiplatelet medicines, and HMG-CoA reductase inhibitors. The patients' comorbidities will also be collected, including the presence of a wound infection, bleeding disorders, sepsis, and whether the surgery was an emergency. Additionally, the history of diabetes, the number of pack-years of smoking, and histories of chronic obstructive pulmonary disease, congestive heart failure, coronary artery disease, chronic kidney disease, and steroid dependence will be documented. Preoperative values of hematocrit, hemoglobin, platelets, creatinine, and albumin will be collected, along with details of the type of anesthesia (general, spinal, or epidural), length of surgery, intraoperative blood loss, postoperative pain ratings, and complications.

Major complications will include pneumonia (as defined by the European Perioperative Clinical Outcome guidelines), myocardial infarction (as defined by the World Health Organization), stroke (defined as a central neurologic deficit persisting postoperatively for more than 24 hours), venous thromboembolism (confirmed on imaging), delirium (confirmed by a psychiatrist), acute kidney injury (as defined by the Kidney Disease: Improving Global Outcomes Criteria), new requirement for dialysis, surgical site infection, and re-operation. Secondary outcomes and mortality will be the primary outcome measures.

Statistical Analysis Descriptive statistics will be employed to summarize the demographic and clinical characteristics of the patients. The association between the type of anesthesia used and postoperative outcomes will be analyzed using the Chi-square test for categorical variables and the Student's t-test for continuous variables. Kaplan-Meier survival analysis will be conducted to estimate survival rates and compare durations of hospital stays between patients receiving different types of anesthesia. Logistic regression will be used to adjust for potential confounders and assess the impact of anesthetic techniques on postoperative complications. Results will be considered statistically significant at a p-value of less than 0.05. All statistical analyses will be performed using the hospital information management system.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with diabetic foot requiring amputation. Patients who underwent toe, ankle, or foot amputation. Patients aged 18 years or older.

Exclusion Criteria:

Patients under the age of 18. Amputations performed for reasons other than diabetic foot. Patients with incomplete or insufficient medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population Description The study population consisted of patients diagnosed with diabetic foot who required amputation and were treated at Ankara Bilkent City Hospital between 2021 and 2023. The population included adults aged 18 years and older, irrespective of sex. This cohort was selected through a retrospective chart review method, ensuring comprehensive inclusion of all eligible patients who underwent toe, ankle, or foot amputations due to diabetic foot during the specified period. The primary focus was on evaluating the outcomes associated with different anesthetic techniques used during these procedures.
  Sampling Method: Non-Probability Sample Minimum Age: 18 Years Maximum Age: Not applicable Sex: All Gender-Based: No Accepts Healthy Volunteers: No
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
30-Day Mortality Rate in Patients Undergoing Diabetic Foot Amputation | Time Frame: 30 days post-surgery.
  This study aims to evaluate the 30-day mortality rate in patients undergoing diabetic foot amputation. Mortality rate is defined as the occurrence of death within 30 days following surgery. The primary focus is to compare the short-term survival effects of different anesthesia techniques (general anesthesia and peripheral nerve block) on these patients.

SECONDARY OUTCOMES:
Composite Morbidity from Potentially Fatal Sequelae | From the date of surgery until hospital discharge, assessed up to 3 months.
  This secondary outcome measure evaluates the occurrence of composite morbidity resulting from potentially fatal sequelae in patients undergoing diabetic foot amputation. This includes major complications such as pneumonia, myocardial infarction, stroke, venous thromboembolism, delirium, acute kidney injury, new requirement for dialysis, surgical site infection, and re-operation. The aim is to assess how different anesthesia techniques impact the rate and severity of these complications.
Hospital Discharge Duration | From the date of surgery until hospital discharge, assessed up to 3 months.
  This secondary outcome measure focuses on the length of hospital stay following diabetic foot amputation. It aims to determine whether the type of anesthesia used (general anesthesia or peripheral nerve block) influences the duration of hospitalization, thereby providing insights into recovery times and healthcare resource utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Semih Başkan, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Semih Başkan, Etimesgut, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Primadhi RA, Septrina R, Hapsari P, Kusumawati M. Amputation in diabetic foot ulcer: A treatment dilemma. World J Orthop. 2023 May 18;14(5):312-318. doi: 10.5312/wjo.v14.i5.312. eCollection 2023 May 18. PMID 37304194
- [Result] Zhu G, Xu J, Dai H, Min D, Guo G. Effect of peripheral nerve block versus general anesthesia on the hemodynamics and prognosis of diabetic patients undergoing diabetic foot Surgery. Diabetol Metab Syndr. 2023 Oct 26;15(1):213. doi: 10.1186/s13098-023-01185-9. PMID 37880794
- [Result] Kim HJ, Park CG, Choi YS, Lee YS, Kwak HJ. Effects of Anesthetic Techniques on the Risk of Postoperative Complications Following Lower Extremity Amputation in Diabetes Patients with Coagulation Abnormalities: A Retrospective Cohort Study Using Propensity Score Analysis. J Clin Med. 2021 Nov 28;10(23):5598. doi: 10.3390/jcm10235598. PMID 34884298